CLINICAL TRIAL: NCT06318130
Title: Comparison of Pacing Lead Design on Left Bundle Branch Pacing Outcomes
Brief Title: Comparison of Pacing Lead Design on Left Bundle Branch Pacing Outcomes: The LEAD_LBBP Randomized Clinical Trial
Acronym: LEAD-LBBP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LEAD-LBBP
Record Dates: First submitted 2024-02-06; First posted 2024-03-19 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Pacemaker DDD
Keywords: Left bundle branch pacing; Lead design; Conduction system pacing

STUDY DESIGN:
Intervention Model Description: A target of 210 participants will be enrolled in this study consisting of two groups and randomised in a 1:1 fashion to either of two groups.
  Group 1: Fixed helix, lumenless pacing lead (FHL) Group 2: Extendable helix, stylet driven pacing lead (EHL)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects will be blinded to the type of pacing lead received. Operators will not be blinded as they will be performing the procedure. Post-procedure, investigators and outcomes assessors will be blinded to the treatment arm during adjudication of outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fixed helix, lumenless pacing lead (FHL) (Active Comparator): Lumenless leads used are fixed helix pacing leads (SelectSecure 3830 pacing lead from Medtronic) during the LBBP procedure.
  Interventions: Device: Fixed helix, lumenless pacing lead.
- Extendable helix, stylet-driven leads (EHL) (Active Comparator): Stylet-driven leads used are extendable helix pacing leads (Biotronik Solia S60 lead from Biotronik or Tendril STS pacing lead from St. Jude Medical) during the LBBP procedure.
  Interventions: Device: Extendable helix, stylet-driven pacing lead.

INTERVENTIONS:
Device: Fixed helix, lumenless pacing lead. — Patients will be randomised to the fixed helix, lumenless pacing lead design during LBBP implantation.
  Arms: Fixed helix, lumenless pacing lead (FHL)
Device: Extendable helix, stylet-driven pacing lead. — Patients will be randomised to the extendable helix, stylet-driven pacing lead design during LBBP implantation.
  Arms: Extendable helix, stylet-driven leads (EHL)

SUMMARY:
This trial seeks to evaluate the performance of the extendable helix, stylet-driven pacing lead (SDL) compared to the fixed helix, lumenless pacing lead (LLL) during left bundle branch pacing (LBBP), with respect to enduring left bundle branch capture on follow-up, incidence of acute lead failure, pacing characteristics including QRS duration, pacing thresholds, R-wave amplitudes and lead impedance, and finally, safety profile during LBBP implantation. These data will guide future lead selection during LBBP implantation in achieving improved procedural success and optimal lead performance.

DETAILED DESCRIPTION:
This study is a single-blind, randomised controlled trial, aimed at evaluating the performance of the extendable helix, stylet driven pacing lead (SDL) compared to the fixed helix, lumenless pacing lead (LLL) during left bundle branch pacing (LBBP). The study is a multicentre study across 3 major hospitals in Singapore, and LBBP performed by independent electrophysiologists experienced in performing LBBP.

The primary objective of the study is to determine differences in incidence of loss of left bundle capture by pacing lead design (LLL vs SDL). The secondary objectives are to determine if lead design affects frequency of lead failure during implantation, investigate differences in short- and medium-term LBBP parameters on follow-up by lead design, and evaluate differences in safety profile between LLL and SDL in LBBP.

This study aims to recruit a target of 210 patients. A previous retrospective study found a loss of LB capture rate of 9% with LLL and 25% with SDL. A sample size of 170 will be required for a type-1 error rate of 5% and power of 80%. Accounting for a dropout rate of 20%, a total of 210 patients will be recruited (105 per group). Eligible subjects will be randomised to either the LLL or the SDL arm. The randomisation list will be generated with a computer-generated sequence in permuted blocks of 4, stratified by centre, to ensure a final allocation ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfil current indications for pacemaker therapy according to international guideline recommendations:

   1. Symptomatic sinus bradycardia/sinus node dysfunction or AV block requiring pacemaker insertion.
   2. Symptomatic heart failure, left ventricular ejection fraction (LVEF) <35%, left bundle branch block and QRS duration >120ms.
   3. Symptomatic heart failure, left ventricular ejection fraction (LVEF) <35%, right bundle branch block and QRS duration >150ms.
   4. LVEF <50% with significant anticipated ventricular pacing requirement of ≥20%.
2. Age ≥21 years old
3. Able to provide informed consent
4. Planned LBBP implantation

Exclusion Criteria:

1. Severe tricuspid regurgitation or previous tricuspid valve intervention requiring implantation of left ventricular lead in the coronary sinus.
2. Unable to provide informed consent.
3. Pregnant women.
4. <21 years of age.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-19 (Estimated); Study Completion 2025-10-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of loss of left bundle branch capture | 12 months
  Loss of LBB capture is defined as the absence of the terminal r/R' complex in V1 during initial threshold interrogations at high pacing outputs and the absence of transitions in paced QRS morphology with decreasing pacing outputs until loss of myocardial capture.

SECONDARY OUTCOMES:
Incidence of acute lead failure | 12 months
  Acute lead failure is defined as defined as structural damage to the pacing lead during implant necessitating the use of a new pacing lead.
Serial changes in pacing thresholds (V) | 12 months
  To compare the differences in pacing thresholds (V) at implant and at 12 months after LBBP implant.
Serial changes in R-wave amplitude (mV) | 12 months
  To compare the differences in R-wave amplitude (mV) at implant and at 12 months after LBBP implant.
Serial changes in lead impedance (ohm) | 12 months
  To compare the differences in lead impedance (ohm) at implant and at 12 months after LBBP implant.
Serial changes in QRS duration (ms) | 12 months
  To compare the differences in QRS duration (ms) at implant and at 12 months after LBBP implant.
Incidence of peri-procedural complications | 12 months
  Complications intraprocedurally and on follow-up will be evaluated, including lead dislodgement, lead fracture during implant, septal perforation, septal vein/arterial injury, pneumothorax, pericardial effusion, wound/pacemaker infection.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Tan, MBBS, Principal Investigator — NUHS
Locations (1):
- National University Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No